CLINICAL TRIAL: NCT03372239
Title: A Phase 1, Randomized Trial to Compare the Oral Bioavailability of Indoximod Salt and Base Formulations and the Effect of Food (Part 1) and to Evaluate the PK and Safety of Single Ascending Doses of Indoximod (Part 2) in Healthy Male Volunteers
Brief Title: Oral Bioavailability,and Food Effect Study and Single Ascending Dose PK Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLG2108
Record Dates: First submitted 2017-12-10; First posted 2017-12-13 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Indoximod
MeSH Terms: interventions — Salts; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Bioavailability and Food Effect (Experimental): Subjects will be randomized to receive the following 3 regimens in randomized sequence:
  1. Single dose of Indoximod base formulation under fasting conditions
  2. Single dose of Indoximod HCL (salt) formulation under fed conditions
  3. Single dose of Indoximod HCL (salt) formulation under fasting conditions
  Interventions: Drug: Indoximod base formulation; Drug: Indoximod HCL (salt) formulation; Other: Placebo
- Part 2: Single Ascending Dose (Experimental)
  Interventions: Drug: Indoximod HCL (salt) formulation; Other: Placebo

INTERVENTIONS:
Drug: Indoximod base formulation — Specified dose on specified days
  Arms: Part 1: Bioavailability and Food Effect
Drug: Indoximod HCL (salt) formulation — Specified dose on specified days
Other: Placebo — Specified dose on specified days

SUMMARY:
This 2-part study will assess the effect of formulation and food on the pharmacokinetics of Indoximod in healthy volunteers. Part 1 is an open-label, 3-period, 6-sequence study. Participants will receive single doses of Indoximod base or salt formulation, in the fasted or fed state. Part 2 is a randomized single ascending dose study of indoximod salt formulation to characterize the PK profile and determine the safety and tolerability of each dose in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18 to 55 years of age, inclusive.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2, and a minimum weight of 50.0 kg.
* Non-smoker for at least 3 months prior to Screening.
* Male subjects with female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception
* Signed and dated written informed consent

Exclusion Criteria:

* History or presence of any clinically significant abnormality, illness, or disease which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or influence the validity of the results of the study.
* Subjects with autoimmune conditions, inflammatory bowel disease, rheumatoid arthritis, and/or subjects who have undergone an organ transplant.
* Self-reported history of substance or alcohol dependence within the past 2 years, and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
* Any medical/surgical procedure or trauma within 4 weeks of the first study drug administration or planned within 1 month of study completion.
* Positive urine drug screen.
* Positive breath alcohol test.
* Evidence of clinically significant hepatic or renal impairment
* Inability to fast for a minimum of 14 hours.
* Inability to swallow large capsules/tablets.
* Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Donation or loss of more than 500 mL whole blood within 1 month preceding entry into the Treatment phase and throughout the study.
* Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
* History of severe allergic reaction (including anaphylaxis) to any substance, or previous status asthmaticus.
* Treatment with an investigational drug within 5 times the elimination half-life, if known (eg, a marketed product), or within 30 days (if the elimination half-life is unknown) prior to first drug administration or is concurrently enrolled in any research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve | up to 20 Days
  Part 1 (Food Effect)
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | up to 20 Days
  Part 1 (Food Effect)
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | up to 4 Days
  Part 2 (Single rising dose)

SECONDARY OUTCOMES:
Percentage of patients with adverse events | up to 34 Days
  Part 1
Percentage of patients with adverse events | up to 16 Days
  Single rising dose

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kennedy, MD, Study Director — NewLink Genetics Inc
Locations (1):
- INC Research/inVentiv Health, Toronto, Ontario, Canada